CLINICAL TRIAL: NCT02202122
Title: Interest of the OSA (Obstructive Sleep Apnea) Predictive Scores in the Prognosis of Postoperative Mortality of Femoral Neck Fractures.
Status: Withdrawn | Type: Observational
Why Stopped: lack of investigators
Sponsor: Astes (Other)
Responsible Party: Principal Investigator, Eric DEFLANDRE, MD, FCCP, Eric DEFLANDRE, MD, FCCP, Astes
Other Study IDs: FNF-OSA
Record Dates: First submitted 2014-07-25; First posted 2014-07-28 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Femoral Neck Fracture
Keywords: Femoral Neck Fractures; Obstructive Sleep Apnea; Perioperative Complications
MeSH Terms: conditions — Femoral Neck Fractures; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Group: OSA Scoring
  Interventions: Other: OSA Scoring

INTERVENTIONS:
Other: OSA Scoring — Comparison of the preoperative OSA scoring (STOP-BANG, DES-OSA, P-SAP and OSA50) with the postoperative mortality at one month.

SUMMARY:
Interest of the four major OSA Predictive Scores (STOP-BANG, P-SAP, DES-OSA, OSA50) in the prognosis of postoperative mortality after femoral neck fracture.

DETAILED DESCRIPTION:
* All patients incoming at the Saint-Luc Bouge Hospital with a femoral neck fracture
* Study between 15/09/2014 and 15/10/2015
* The four OSA predictive scores will be collected
* Evaluation of mortality at 1 month

ELIGIBILITY:
Inclusion Criteria:

* All patients with femoral neck fractures
* Incoming at the Saint-Luc Bouge Hospital
* Between 15/09/2014 and 15/10/2015

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with femoral neck fractures
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Impact OSA predictive scores on mortality prognosis | 1 month
  Impact of the four major OSA predictive scores (STOP-BANG, P-SAP, OSA50 et DES-OSA) on the mortality prognosis after surgery for femoral neck fracture

CONTACTS AND LOCATIONS:
Overall Officials: Eric P Deflandre, MD, FCCP, Principal Investigator — Astes
Locations (1):
- Clinique Saint-Luc de Bouge, Namur, Namur, Belgium